CLINICAL TRIAL: NCT05701865
Title: Biphasic Effects of Acute Alcohol Intoxication on Bystander Intervention for Sexual Violence
Brief Title: Biphasic Effects of Acute Alcohol Intoxication on Bystander Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Ruschelle Leone, Assistant Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R21AA029225 (NIH)
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol Intoxication (Experimental): Participant will receive alcohol, the dose of which will be administered to result in a breath alcohol concentration of .08%.
  Interventions: Behavioral: Alcohol Intoxication- Ascending Limb; Behavioral: Alcohol Intoxication- Descending Limb
- No-Alcohol Control (Active Comparator): Participant will receive a no alcohol control beverage, therefore their breath alcohol concentration will be .00%.
  Interventions: Behavioral: No Alcohol Control

INTERVENTIONS:
Behavioral: Alcohol Intoxication- Ascending Limb — Participants will be assigned to moderate alcohol dose condition (target breath alcohol concentration .08%) with NIAAA approved alcohol administration procedures and complete the study task on the ascending limb
  Arms: Alcohol Intoxication
Behavioral: Alcohol Intoxication- Descending Limb — Participants will be assigned to moderate alcohol dose condition (target breath alcohol concentration .08%) with NIAAA approved alcohol administration procedures and complete the study task on the descending limb
  Arms: Alcohol Intoxication
Behavioral: No Alcohol Control — Participants will be assigned to a no alcohol control condition
  Arms: No-Alcohol Control

SUMMARY:
The goal of this experimental study is to examine the effect of alcohol, gender, and bystander attitudes on bystander barriers and sexual violence intervention among young adult men and women (age 21-20). The main questions it aims to answer are:

* Does alcohol intoxication and gender influence bystander barriers and sexual violence intervention?
* Does alcohol intoxication have a greater impact on bystander barriers and sexual violence intervention among men, compared to women?
* Does alcohol intoxication have a greater impact on bystander barriers and sexual violence intervention among those with higher, compared to lower, prosocial bystander attitudes?

Participants will be randomly assigned to one of two beverage conditions (alcohol or control beverage) and those assigned to alcohol will complete the study on either the ascending or descending alcohol limb. Participants will project themselves into a heat-of-the moment, risky sexual violence scenario that will assess bystander barriers and behavioral intentions. Researchers will compare those assigned to the alcohol and control beverage condition and men/women to see if this impacts bystander barriers and sexual violence intervention.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21 and 30
* Report that on at least 3 days in the past year they have consumed an alcohol quantity on a single occasion that was equal or greater to the dose administered in the lab

Exclusion Criteria:

* Currently seeking treatment or in recovery for an alcohol or substance use disorder
* A medical condition or medication use in which alcohol consumption is medically contraindicated
* Pregnant, nursing, or has engaged in sexual intercourse without effective contraception in the past two weeks
* If the participant is less than six feet tall and weighs over 250 pounds or is over six feet tall and weighs over 300 pounds

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Man or woman
Enrollment: 192 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Articulated Thoughts of Barriers to Bystander Intervention | 35 minutes to 2.5 hours post-drinking
  Participants will verbally respond to a heat-of-the-moment scenario where they are a bystander of a risky alcohol-related sexual violence situation using the articulate thoughts in simulated situations paradigm [Davidson et al., 1983].
Articulated Thoughts of Intentions to Intervene as a Bystander | 35 minutes to 2.5 hours post-drinking
  Participants will verbally respond to a heat-of-the-moment scenario where they are a bystander of a risky alcohol-related sexual violence situation using the articulate thoughts in simulated situations paradigm [Davidson et al., 1983]

CONTACTS AND LOCATIONS:
Overall Officials: Ruschelle M Leone, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available in the NIAAA Data Archive.

DOCUMENTS (1):
  • Informed Consent Form (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT05701865/ICF_000.pdf